CLINICAL TRIAL: NCT00334646
Title: An Open Label, Repeat Dose, Randomized, Two Period Crossover Study to Investigate the Potential Pharmacokinetic Interactions Between Oral GW679769 and Intravenous Cyclophosphamide in Cancer Patients
Brief Title: Cyclophosphamide Drug Interaction Study In Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: compound terminated
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NKV103444
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: cyclophosphamide; CINV; Chemotherapy induced nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Cyclophosphamide

ARMS (2):
- Arm A (Experimental): cyclophosphamide + dexamethasone + ondansetron
  Interventions: Drug: IV Cyclophosphamide 500-700mg/m2
- Arm B (Experimental): cyclophosphamide + dexamethasone + ondansetron + GW679769
  Interventions: Drug: Oral GW679769

INTERVENTIONS:
Drug: Oral GW679769 — 150mg oral, once daily on days 1-3
  Arms: Arm B
Drug: IV Cyclophosphamide 500-700mg/m2 — IV Cyclophosphamide 500-700mg/m2 on day 1 of each cycle
  Other Names: Oral GW679769
  Arms: Arm A

SUMMARY:
This study is designed to evaluate the potential pharmacokinetic interaction between oral GW679769 and IV (intravenous) cyclophosphamide when administered to cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of cancer.
* Undergoing chemotherapy with a cyclophosphamide regimen with a cyclophosphamide dose of 500 - 700 mg/m2 and a cycle duration of 14-28 days.
* Adequate hematologic, renal and hepatic function.

Exclusion Criteria:

* Pregnant or lactating.
* CNS (central nervous system) metastases.
* Active systemic infection or any other poorly controlled medical condition.
* Patients cannot take CYP3A4 inhibitors within 7 days of study treatment or CYP3A4 inducers within 48 days of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-08-10 (Actual); Primary Completion 2009-10-14 (Actual); Study Completion 2009-10-14 (Actual)

PRIMARY OUTCOMES:
Cmax and AUC of cyclophosphamide and 4-hydroxycyclophosphamideSafety and tolerability parameters including pharmacoeconomics, blood pressure, heart rate, ECG, laboratory tests, clinical observation and adverse event reporting. | throughout the study

SECONDARY OUTCOMES:
Terminal t1/2, Vd, and Cl of cyclophosphamideTerminal t1/2 of 4-hydroxycyclophosphamideAUC ratio of 4-hydroxycyclophosphamide and cyclophosphamideANC nadir | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (3):
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, The Bronx, New York
- GSK Investigational Site, Christchurch, New Zealand
- GSK Investigational Site, Lund, Sweden

REFERENCES:
- See also: Results for study NKV103444 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/NKV103444?search=study&study_ids=NKV103444#rs